CLINICAL TRIAL: NCT05553847
Title: Automated Oxygen Titration to Improve Activities of Daily Living in Patients With Chronic Obstructive Pulmonary Disease on Home Oxygen
Brief Title: Automated Oxygen Titration in Daily Life in Patients With COPD on Home Oxygen
Acronym: DaiLiHOT_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Örebro University, Sweden (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Linette Marie Kofod, Physiotherapist, Primary investigator, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Fys1977
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Activity; Automated oxygen titration; ADL; long term oxygen treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: multicentre double blinded randomized crossover trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded for the oxygen supply. An independent person will prepare the oxygen setup with usual fixed dose or automated titration. The setup i covered. The assessor conducting the tests is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual oxygen dose (No Intervention): A Glittre-ADL tests will be performed and the patients will use their usual fixed dose of oxygen. Pulse rate and saturation will continuously be registered during the test. Before, and after the Glittre-ADL, the patients will be asked the rate their level of dyspnea using Borg Dyspnea Scale
- Automated oxygen dose (Experimental): A Glittre-ADL tests will be performed and the patients will use automated oxygen titration set at an SpO2-target of 90 to 94 % and an oxygen flow of 0 - 8 liters/min. Pulse rate, oxygen flow rate and saturation will continuously be registered during the test. Before, and after the Glittre-ADL, the patients will be asked the rate their level of dyspnea using Borg Dyspnea Scale
  Interventions: Other: Automated oxygen titration based on the oxygen saturation during activity

INTERVENTIONS:
Other: Automated oxygen titration based on the oxygen saturation during activity — A device will be used, which automatically adjusts the oxygen flow to the dosage necessary for keeping the saturation at the recommended level (90-94%). If the saturation falls below 90%, oxygen flow will increase, and if the saturation increases above 94%, oxygen flow decreases in order to stay on target.
  Arms: Automated oxygen dose

SUMMARY:
The purpose of this study is to examine the effect of automated oxygen titration compared to the usual fixed dose oxygen on the patient's ability to perform activities of daily living.

DETAILED DESCRIPTION:
The patient's ability to perform ADL assessed by the Glittre-ADL test with automatic oxygen titration compared to usual fixed dose will be examined.

The patients will be invited to a visit at one of the participating hospitals. The Glittre-ADL will be performed according to the protocol validated by Skumlien et al. The first test is performed for familiarization in order to avoid a learning effect in the primary tests. The patients will use the fixed-dose oxygen, established after titration to a SpO2 of 90-94 % at rest.

After the familiarization test and gathering of demographics, further two Glittre-ADL tests will be performed on the same day or at another day pending on patient preference. In random order the patients will use A) automated oxygen titration set at an SpO2-target of 90 to 94 % and an oxygen flow of 0 - 8 liters/min and B) their usual fixed dose of oxygen. In both arms O2matic will monitor pulse rate and saturation continuously during the test, but only in the automated oxygen therapy arm O2matic adjusts the oxygen flow. The patients will all use a rollator as walking aid. The oxygen equipment will be placed in the rollator and the tests will be conducted without the steps (due to the use of rollator). The minimum interval between tests will be 20 minutes or until the vital values and symptoms are returned to baseline. Before, and after the Glittre-ADL, the patients will be asked the rate their level of dyspnea using Borg Dyspnea Scale.

Study Analysis Plan

1. Paired sample t-test: time used in the Glittre test using AutOx vs Time used using Fixed oxygen (in seconds)
2. Paired sample t-test: Borg score after Glittre using Autox vs Borg score after Glittre when using Fixed oxygen (on a scale from 0-10) A test for carryover effect will be performed by comparing the first and the second tests before being divided into the Autox and fixed oxygen groups.

Variables will be examined for normality and analyzed with either a paired t-test (in case of normality) or Wilcoxon-signed-rank test (in case of non-normality). The median of the differences between tests will be used for a value. The number of patients who reach a Minimal Clinically Important Difference (MCID) in either the Dyspnea score or in time used in the Glittre test will be reported.

Difference in time spent within saturation intervals will be extracted from the CSV files and combined using Excel.

IBM SPSS Statistics for Windows, ver. 29.0.1.0 will be used for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Verified history of COPD with FEV1/FVC < 0.70 and FEV1 < 50 %
* Hypoxemic at rest (SpO2≤ 90 %) and fulfilment of general national criteria for LTOT

  * Partial pressure of Oxygen (PaO2) (without oxygen supplement) ≤7.3 kPa in clinically stable and optimally treated condition
  * Increase in PaO2 after oxygen supplementation (to 8.0-9.0 kPa) without decrease in arterial pH (> 0.03 kPa)
  * The oxygen is used at least 15 hours daily (optimally 24 hours daily)
  * The treatment is handled by hospital departments with lung medical expertise.
* Able to walk at least 30 meters
* Age >18, Cognitively able to participate in the study and willing to give informed consent

Exclusion Criteria:

* Pulmonary or cardiac condition other than COPD limiting physical performance
* Unstable heart condition or stenotic aortic valve disease
* A physical condition including paralysis, lower extremity pain, or back problem limiting physical performance
* Exacerbation in COPD treated with either antibiotics or prednisolone within the last 3 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Time used for the Glittre-ADL test | Immediately after intervention (control arm test and automated oxygen titration arm) on the same day
  Change in time used to complete the Glittre-ADL test with automated titration compared to fixed-dose treatment

SECONDARY OUTCOMES:
Dyspnea | Immediately after the intervention
  Change in Dyspnea Borg (in units from 0-10) scores after performing Glittre ADL test between arms
Saturation | Immediately after the intervention
  Change in time spent within acceptable SpO2-interval (SpO2 90 - 94 %) and time spent with moderate hypoxemia (SpO2 < 88 %) and severe hypoxemia (SpO2 < 85 %) in the two Glittre-ADL tests
Oxygen consumption | Immediately after the intervention
  Change in average oxygen consumption between the two tests

CONTACTS AND LOCATIONS:
Overall Officials: Linette M Kofod, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data could be available on reasonable request, but needs to follow the rules set by the danish Data Protection Agency.

REFERENCES:
- [Derived] Kofod LM, Hansen EF, Brocki BC, Kristensen MT, Roberts NB, Westerdahl E. Optimised oxygenation improves functional capacity during daily activities in patients with COPD on long-term oxygen therapy: a randomised crossover trial. Thorax. 2025 Oct 15;80(11):803-809. doi: 10.1136/thorax-2024-221883. PMID 40473413